CLINICAL TRIAL: NCT00749671
Title: To Assess the Utility of BIS Monitoring in the Administration of Moderate Sedation in Patients Undergoing Implantable Cardioverter -Defibrillator (ICD) Implantation With Defibrillatory Threshold (DFT) Testing
Brief Title: Bispectral Index Monitoring During Testing in the Electrophysiology Lab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, James Cook, Director, EP Lab, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-186
Record Dates: First submitted 2007-11-13; First posted 2008-09-09 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Tachycardia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICD testing BIS (Active Comparator): Bispectral Index Monitoring will be used to assess adequacy of moderate sedation during DFT.
  Interventions: Device: Bispectral index monitoring
- ICD testing Ramsey (Active Comparator): Ramsey Sedation Scale will be used to assess adequacy of moderate sedation during DFT
  Interventions: Other: Ramsey Sedation Scale

INTERVENTIONS:
Device: Bispectral index monitoring — The monitoring of the EEG signal is designed to determine if the sedation is adequate.
  Arms: ICD testing BIS
Other: Ramsey Sedation Scale — The determination of the degree of sedation is accomplished using an established sedation scale.
  Arms: ICD testing Ramsey

SUMMARY:
BACKGROUND Physician-guided moderate sedation, administered by a Registered Nurse has been the standard of practice for patients undergoing a wide range of electrophysiology procedures during the past decade. Currently a subjective sedation assessment tool is the standard of practice within the Electrophysiology Lab (EP Lab). Bispectral Index monitoring (BIS) is an objective measure of the depth of sedation presently employed at Baystate Medical Center in the Intensive Care Unit and within the department of anesthesia.

AIM The aim of this research study is to assess the utility of BIS monitoring in measuring the depth of sedation in patients undergoing defibrillation threshold testing (DFT). Our primary endpoint is: A change in OAAS scores of one point at the 30 minute data collection time period.

Our secondary endpoints are: Lack of explicit recall of DFT testing and measurement of perioperative level of comfort.

STUDY DESIGN AND SCOPE The population to be studied is those patients receiving a primary ICD implant or an ICD battery change with defibrillation threshold testing (DFT).

All patients who have consented for ICD placement and DFT testing with moderate sedation will be invited to participate in this research study. Patients who are not candidates for DFT testing, as is determined by the EP physician, will be excluded from the study.

Demographic data including: age, gender, BMI, current medications and history of sleep apnea will be collected. Data detailing the amount of drug administered during the procedure and any use of reversal agents, will be retrieved from the medical record.

The study will be conducted within the Electrophysiology lab at Baystate Medical Center. An enrollment of 60 subjects is expected to be completed within 6 months. 30 patients will originate from the outpatient population and 30 from the inpatient.

Follow up assessments using the OAAS scale will be completed at 30 min, 1 hour and 4 hours post procedure. Also, perioperative comfort and recall of DFT testing will be assessed at the 4 hour mark.

DETAILED DESCRIPTION:
BACKGROUND Physician-guided moderate sedation, administered by a Registered Nurse has been the standard of practice for patients undergoing a wide range of electrophysiology procedures during the past decade. Currently a subjective sedation assessment tool is the standard of practice within the Electrophysiology Lab (EP Lab). Bispectral Index monitoring (BIS) is an objective measure of the depth of sedation presently employed at Baystate Medical Center in the Intensive Care Unit and within the department of anesthesia.

AIM The aim of this research study is to assess the utility of BIS monitoring in measuring the depth of sedation in patients undergoing defibrillation threshold testing (DFT). Our primary endpoint is: A change in Observer's Assessment of Alertness/Sedation Scales (OAAS) scores of one point at the 30 minute data collection time period.

Our secondary endpoints are: Lack of explicit recall of DFT testing and measurement of perioperative level of comfort.

STUDY DESIGN AND SCOPE The population to be studied is those patients receiving a primary ICD implant or an ICD battery change with defibrillation threshold testing (DFT).

All patients who have consented for ICD placement and DFT testing with moderate sedation will be invited to participate in this research study. Patients who are not candidates for DFT testing, as is determined by the EP physician, will be excluded from the study.

Demographic data including: age, gender, BMI, current medications and history of sleep apnea will be collected. Data detailing the amount of drug administered during the procedure and any use of reversal agents, will be retrieved from the medical record.

The study will be conducted within the Electrophysiology lab at Baystate Medical Center. An enrollment of 60 subjects is expected to be completed within 6 months. 30 patients will originate from the outpatient population and 30 from the inpatient.

Follow up assessments using the OAAS scale will be completed at 30 min, 1 hour and 4 hours post procedure. Also, perioperative comfort and recall of DFT testing will be assessed at the 4 hour mark.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are having ICD placement and DFT testing will be invited to participate in this research study.

Exclusion Criteria:

* Patients who are not candidates for DFT testing, as is determined by the EP physician
* An example of such a patient would be one who is hemodynamically unstable;
* DFT testing is contraindicated in this case.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: james cook, md, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bispectral Index Monitoring: Bispectral index monitoring using Aspect Monitor: The monitoring of the EEG signal is designed to determine if the sedation is adequate.
- Ramsey Scale Monitoring: Group assigned to sedation monitoring using the Ramsey Scale for ICD testing
Period: Overall Study
Arm/Group | Bispectral Index Monitoring | Ramsey Scale Monitoring
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ICD Testingwith Bispectral Monitoring: Bispectral Index Monitoring
  Bispectral index monitoring using Aspect Monitor: The monitoring of the EEG signal is designed to determine if the sedation is adequate.
- Nurse Administered Moderate Sedation: Moderate sedation using the Ramsey scale as assessed by a nurse trained and dedicated to monitoring the patient
- Total: Total of all reporting groups
Arm/Group | ICD Testingwith Bispectral Monitoring | Nurse Administered Moderate Sedation | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — While gender was recorded at baseline, we no longer have access to the dataset to tabulate
  Participants
    Female | NA — dataset not accessible | NA — dataset not accessible | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — dataset not accessible | NA — dataset not accessible | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Observer's Assessment of Alertness/Sedation (OAAS) Rating Scale at 30 Minutes
Description: Sedation level was evaluated and graded according to the observer's assessment of alertness/sedation (OAAS) rating scale. This scale has 6 possible measures of consciousness:
  OAAS score 5-awake and responds readily to name spoken in normal tone.
  OAAS score 4-lethargic responses to name in normal tone.
  OAAS score 3-responds only after name is called loudly and/or repeatedly.
  OAAS score 2-responds only after name called loudly and mild shaking.
  OAAS score 1-does not respond when name is called loudly and mild shaking or prodding.
  OAAS score 0-does not respond to noxious stimulation.
Time Frame: 30 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- ICD Testing: Bispectral Index Monitoring
  Bispectral index monitoring using Aspect Monitor: The monitoring of the EEG signal is designed to determine if the sedation is adequate.
- ICD testing2: Ramsey Sedation Scale
  Ramsey Sedation Scale: The determination of the degree of sedation is accomplished using an established sedation scale.
Arm/Group | ICD Testing | ICD testing2
Number analyzed (Participants) | 11 | 9
units on a scale | 4.27 [3.35 to 5.19] | 4.33 [3.33 to 5.33]

2. Secondary Outcome: Patient Recall of Defibrillation Testing
Description: The patient recall of the testing will be assessed at 30 minutes, as answered with a yes/no.
Time Frame: 30 minutes
Measure: Number; unit: percentage of patients with DFT recall
Arm/Group | ICD Testing BIS | ICD Testing Ramsey
Number analyzed (Participants) | 11 | 9
percentage of patients with DFT recall | 0 | 0

ADVERSE EVENTS:
Arm/Group | ICD Testingwith Bispectral Monitoring | Nurse Administered Moderate Sedation
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No